CLINICAL TRIAL: NCT01901835
Title: The Effects of a Media Diversion on Quality of Life in Patients Receiving Chemotherapy for Recurrent Gynecologic Cancers
Brief Title: Media Diversion in Improving Quality of Life in Patients With Recurrent Gynecologic Cancers Receiving Chemotherapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Supportive Care
Other Study IDs: UW13037; NCI-2013-01284 (Registry Identifier: NCI Trial ID); 2013-0618 (Other: Institutional Review Board); P30CA014520 (NIH); A532820 (Other: UW Madison); SMPH/OBSTET & GYNECOL/ (Other: UW Madison)
Record Dates: First submitted 2013-07-12; First posted 2013-07-17 (Estimated); Last update posted 2019-11-19 (Actual); Status verified 2017-03

CONDITIONS: Female Reproductive Cancer
MeSH Terms: interventions — Mind-Body Therapies

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I (humorous followed by non-humorous movies) (Experimental): Participants are provided headphones and a tablet and choose among a selection of humorous movies. Upon the third course of chemotherapy, participants are provided a selection of non-humorous movies.
  Interventions: Procedure: mind-body intervention procedure; Other: survey administration; Procedure: quality-of-life assessment
- Arm II (non-humorous followed by humorous movies) (Experimental): Participants are provided headphones and a tablet and choose among a selection of non-humorous movies. Upon the third course of chemotherapy, participants are provided a selection of humorous movies.
  Interventions: Procedure: mind-body intervention procedure; Other: survey administration; Procedure: quality-of-life assessment

INTERVENTIONS:
Procedure: mind-body intervention procedure — Participate in media diversion with humorous and non-humorous movies
  Other Names: mind-body interventions
Other: survey administration — Ancillary studies
Procedure: quality-of-life assessment — Ancillary studies
  Other Names: quality of life assessment

SUMMARY:
This randomized clinical trial studies media diversion in improving quality of life in patients with recurrent gynecologic cancers receiving chemotherapy. Media diversion may improve mood and quality of life in patients having cancer treatment.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To analyze the impact of a media-based intervention on patient mood during the receipt of chemotherapy for recurrent gynecologic cancers.

OUTLINE: are randomized to 1 of 2 arms.

ARM I: Participants are provided headphones and a tablet and choose among a selection of humorous movies. Upon the third course of chemotherapy, participants are provided a selection of non-humorous movies.

ARM II: Participants are provided headphones and a tablet and choose among a selection of non-humorous movies. Upon the third course of chemotherapy, participants are provided a selection of humorous movies.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with pathologically-proven gynecologic malignancies
* Subjects who have previously completed primary treatment for a gynecologic malignancy
* Patients receiving chemotherapy for a recurrent gynecologic cancer at the University of Wisconsin-Madison Carbone Cancer Center (UWCCC)
* Patients must be English speaking
* Patients must have the ability to use audio media and read and understand written English

Exclusion Criteria:

* Patients unable to use audio or video media due to auditory or ocular dysfunction
* Patients unable to read written English
* Patients who are prisoners or incarcerated

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2014-02-12; Primary Completion 2016-05-24 (Actual); Study Completion 2017-02-08 (Actual)

PRIMARY OUTCOMES:
Patient-reported mood using the Positive and Negative Affect Scale-Expanded Form (PANAS-X) instrument | Up to day 1 of course 3 of chemotherapy
  Summarized in terms of means, standard deviations and ranges, stratified by group and assessment time point. Absolute and percentage changes from baseline within each group will be calculated and reported in terms of means and the corresponding 95% confidence intervals. Changes from baseline will be evaluated using a paired t-test. A Grizzle model for a 2 X 2 cross-over design will be used to compare changes in PANAS-X positive and negative affect scores between groups.

SECONDARY OUTCOMES:
Humor Styles Questionnaire (HSQ) total score | Up to day 1 of course 3 of chemotherapy
  Summarized in terms of means, standard deviations and ranges, stratified by group and assessment time point. Absolute and percentage changes from baseline within each group will be calculated and reported in terms of means and the corresponding 95% confidence intervals. Changes from baseline will be evaluated using a paired t-test. A Grizzle model for a 2 X 2 cross-over design will be used to compare changes in HSQ total scores between groups.
Brief Fatigue Inventory (BFI) total score | Up to day 1 of course 3 of chemotherapy
  Summarized in terms of means, standard deviations and ranges, stratified by group and assessment time point. Absolute and percentage changes from baseline within each group will be calculated and reported in terms of means and the corresponding 95% confidence intervals. Changes from baseline will be evaluated using a paired t-test. A Grizzle model for a 2 X 2 cross-over design will be used to compare changes in BFI total scores between groups.
Ease of use (EoS) score | Up to day 1 of course 3 of chemotherapy
  Assessed with a Likert scale at the completion of the subject's participation to understand how the intervention may be improved should results of this study favor implementation into standard clinical procedure for future patients. Summarized in terms of medians and ranges, stratified by group and assessment time point. Changes from baseline within each group will be evaluated using a nonparametric Wilcoxon Signed Rank test
Quality of materials (QOM) score | Up to day 1 of course 3 of chemotherapy
  Assessed with a Likert scale at the completion of the subject's participation to understand how the intervention may be improved should results of this study favor implementation into standard clinical procedure for future patients. Summarized in terms of medians and ranges, stratified by group and assessment time point. Changes from baseline within each group will be evaluated using a nonparametric Wilcoxon Signed Rank test

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Rose, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin Hospital and Clinics, Madison, Wisconsin, United States

REFERENCES:
- See also: University of Wisconsin Carbone Cancer Center — https://cancer.wisc.edu/